CLINICAL TRIAL: NCT02354976
Title: A Double-blind Randomized Placebo-controlled, Parallel-group 12 Week Study to Investigate the Effects of Epanova® Compared to Placebo and Compared to Fenofibrate on Liver Fat Content in Hypertriglyceridemic overwEight subjeCTs; EFFECT I
Brief Title: A Double-blind Randomized Placebo-controlled Study Comparing Epanova and Fenofibrate on Liver Fat in Overweight Subjects.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5881C00007
Record Dates: First submitted 2015-01-30; First posted 2015-02-03 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD; Hypertriglyceridemia
Keywords: omega-3 carboxylic acid
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Hypertriglyceridemia | interventions — omega-3 carboxylic acid; Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Omega-3 carboxylic acids 4g / day (Experimental)
  Interventions: Drug: Omega-3 carboxylic acid
- Fenofibrate 200mg (Active Comparator)
  Interventions: Drug: Fenofibrate 200mg

INTERVENTIONS:
Drug: Placebo — Placebo matching to Omega-3 carboxylic acids (olive oil)
  Arms: Placebo
Drug: Omega-3 carboxylic acid — 4 g administered as 4 x 1 g capsules
  Arms: Omega-3 carboxylic acids 4g / day
Drug: Fenofibrate 200mg — 200mg capsule administered once daily
  Arms: Fenofibrate 200mg
Drug: Placebo — Placebo matching to fenofibrate 200mg
  Arms: Placebo

SUMMARY:
This study is a double-blind randomized, placebo-controlled, parallel-group, 12 week study performed in 2 centres in Sweden to assess the effect of Omega-3 carboxylic acids and fenofibrate on liver fat measured with magnetic resonance imaging (MRI) in patients with over-weight and hypertriglyceridemia.

ELIGIBILITY:
Inclusion Criteria: - Provision of informed consent

* Men or women ≥40 years and ≤75 years with suitable veins for cannulation or repeated venepuncture
* Have serum triglycerides ≥1.7 mM
* Have liver fat content as assessed by MRI >5.5%
* Have a body mass index (BMI) >25 and ≤40 kg/m2

  , Exclusion Criteria: - History of or presence of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* Creatinine clearance <60 mL/min at screening (Cockcroft-Gault formula).
* Severe hepatic insufficiency and/or significant abnormal liver function defined as aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >3x ULN
* Total bilirubin >2.0 mg/dL (34.2 µmol/L)
* Type 2 diabetes, as defined by WHO criteria e.g. fasting plasma Glucose >7.0 mM or use of antidiabetic therapy
* Any clinically significant abnormalities in clinical chemistry, haematology or urinalysis results as judged by the investigator. This includes signs of liver disease other than NAFLD that motivates further investigations of treatment based on clinical judgement
* Recent history (past 12 months) of drug abuse or alcohol abuse. Alcohol abuse was to be defined as >14 drinks per week (1 drink = 35 cl beer, 14 cl wine, or 4 cl hard liquor) or as judged by the investigator

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2016-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lind, Professor, Principal Investigator — Uppsala University Hospital. Uppsala Sweden
Locations (4):
- Sweden (4):
  - Research Site, Gothenburg
  - Research Site, Malmo
  - Research Site, Stockholm
  - Research Site, Uppsala

REFERENCES:
- [Derived] Oscarsson J, Onnerhag K, Riserus U, Sunden M, Johansson L, Jansson PA, Moris L, Nilsson PM, Eriksson JW, Lind L. Effects of free omega-3 carboxylic acids and fenofibrate on liver fat content in patients with hypertriglyceridemia and non-alcoholic fatty liver disease: A double-blind, randomized, placebo-controlled study. J Clin Lipidol. 2018 Nov-Dec;12(6):1390-1403.e4. doi: 10.1016/j.jacl.2018.08.003. Epub 2018 Aug 10. PMID 30197273

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 4 centers in Sweden between 01 September 2015 and 26 May 2016.
Pre-assignment Details: The study duration was up to 15 weeks, consisting of an initial screening period lasting up to 2 weeks, a 12-week treatment period, and a follow-up telephone call within 1 week after the last dose of study drug. A total of 78 subjects were randomized.
Groups:
- Epanova: Epanova 4 g/day + placebo to Fenofibrate
- Fenofibrate: Fenofibrate 200 mg/ day + placebo to Epanova
- Placebo: Placebo to Epanova + placebo to Fenofibrate
Period: Overall Study
Arm/Group | Epanova | Fenofibrate | Placebo
Started | 25 | 27 | 26
Completed | 23 | 26 | 23
Not Completed | 2 | 1 | 3
Not completed — Other - reason not specified | 1 | 0 | 1
Not completed — Study-specifc withdrawal criteria | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epanova | Fenofibrate | Placebo | Total
Number analyzed (Participants) | 25 | 27 | 26 | 78
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.0 (7.79) [44 to 74] | 61.7 (7.78) [46 to 74] | 60.8 (7.85) [45 to 72] | 60.8 (7.73) [44 to 74]
Age, Customized [Count of Participants; unit: Participants]
  <50 | 3 | 3 | 1 | 7
  >=50 - <65 | 16 | 14 | 15 | 45
  >=65 | 6 | 10 | 10 | 26
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 9 | 12 | 12 | 33
  Male | 16 | 15 | 14 | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 0 | 2
  Other | 1 | 0 | 0 | 1
  White | 23 | 26 | 26 | 75

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Ratio (Week 12/Baseline) of % Liver Fat as Assessed by MRI (Epanova Versus Placebo)
Description: To evaluate the efficacy of Epanova compared to placebo with respect to reduction in liver fat content (%) at the end of 12 weeks of double-blinded treatment.
Time Frame: Baseline and 12 weeks
Population: The Full Analysis Set included all randomized patients, regardless of whether they took study medication or not. In this set, patients were analyzed according to their randomized treatment assignment.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio of % liver fat
Arm/Group | Epanova | Placebo
Number analyzed (Participants) | 22 | 23
ratio of % liver fat | 0.98 [0.82 to 1.17] | 1.04 [0.95 to 1.13]
Statistical Analysis 1: Comparison: Epanova vs Placebo; Test type: Other; p = 0.407, Mixed Models Analysis; Geometric mean ratio for difference = 0.92, 95% CI 2-sided [0.76 to 1.12]

2. Secondary Outcome: Geometric Mean Ratio (Week 12/Baseline) of % Liver Fat as Assessed by MRI (Epanova Versus Fenofibrate)
Description: To evaluate the efficacy of Epanova compared to Fenofibrate with respect to reduction in liver fat content (%) at the end of 12 weeks of double-blinded treatment.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio of % liver fat
Arm/Group | Epanova | Fenofibrate
Number analyzed (Participants) | 22 | 26
ratio of % liver fat | 0.98 [0.82 to 1.17] | 1.17 [0.99 to 1.37]
Statistical Analysis 1: Comparison: Epanova vs Fenofibrate; Test type: Other; p = 0.077, Mixed Models Analysis; Geometric mean ratio for difference = 0.84, 95% CI 2-sided [0.70 to 1.02]

ADVERSE EVENTS:
Arm/Group | Epanova | Fenofibrate | Placebo
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 17/25 | 15/27 | 8/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epanova (N=25) | Fenofibrate (N=27) | Placebo (N=26)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epanova (N=25) | Fenofibrate (N=27) | Placebo (N=26)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 2 (2) | 4 (4)
Flatulence (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder pain (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Petachiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tendon operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No